CLINICAL TRIAL: NCT04825665
Title: The Effect of Two Different Types of Forces on Possible Root Resorption in Relation to Dentin Phosphoprotein Levels: A Randomized Controlled Clinical Trial
Brief Title: The Effect of Two Different Types of Forces on Possible Root Resorption in Relation to Dentin Phosphoprotein Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sherifa Ghaleb (Other)
Responsible Party: Sponsor-Investigator, Sherifa Ghaleb, Instructor, Principal investigator, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Dentin Phosphoprotein
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Root Resorption
Keywords: Root resorption; Gingival crevicular fluid; Dentin Phosphoprotein; Continuous force; Intermittent force
MeSH Terms: conditions — Root Resorption

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous force (Experimental): A buccally directed continuous tipping force of 150 g is applied to the maxillary first premolar on one side
  Interventions: Other: Continuous force
- Intermittent force (Experimental): A buccally directed tipping force of 150 g removed every 21 days for a 7-day rest period applied to the maxillary first premolar on one side
  Interventions: Other: Intermittent force

INTERVENTIONS:
Other: Continuous force — A buccally directed continuous tipping force of 150 g is applied to the maxillary first premolar by a cantilever spring made of 0.017" x 0.025" beta-titanium-molybdenum alloy inserted in the tube of the upper first molar, bypassing the second premolar and attaching to the upper first premolar. The buccal tipping force will be checked and reactivated to the original level on the 28th day of the 8 week study period.
  Arms: Continuous force
Other: Intermittent force — A buccally directed tipping force of 150 g is applied to the maxillary first premolar by a cantilever spring made of 0.017" x 0.025" beta-titanium-molybdenum alloy inserted in the tube of the upper first molar and attaching to the upper first premolar. The buccal tipping force will be removed every 21 days for a 7-day rest period, where a passive wire of the same gauge and material of the cantilever spring (0.017" x 0.025" beta-titanium-molybdenum alloy) will be placed instead to maintain the position of the upper first premolar during the rest period.
  Arms: Intermittent force

SUMMARY:
External root resorption is a common unfavourable sequel of orthodontic treatment. Although diagnosis of root resorption is usually done by radiographs; they are technique sensitive. Dentine phosphoprotein, a non-collagenous protein, is suggested to be released into the gingival crevicular fluid during active root resorption, serving as a good diagnostic tool. Also, the manner of force application is a modifiable factor suggested to affect root resorption.

DETAILED DESCRIPTION:
Early detection of teeth at risk of severe resorption is crucial.At present, using radiographs is common but detecting only resorption after 60-70% of the mineralized tissue is already lost. Moreover, they only provide two-dimensional information, identifying apical change primarily. Also, radiographs cannot indicate if the process of root resorption is still active for monitoring its progress and additional radiation exposure to the patient will be needed. Therefore, a safer, more reliable alternative method to clinically diagnose early stages of root resorption is needed and may include detecting biomarkers in gingival crevicular fluid. Furthermore, the relationship between the manner of orthodontic force application and orthodontically induced root resorption is under study. It has been suggested that pausing orthodontic forces during treatment may reduce the amount of root resorption, likely due to cementum repair during the inactive period. This is important specifically in individuals who are biologically and genetically prone to root resorption. The aim of the study is to compare the extent of root resorption between controlled continuous and intermittent orthodontic forces using levels of dentin phosphoprotein in gingival crevicular fluid.

ELIGIBILITY:
Inclusion Criteria:

* Malocclusion that requires extraction of first maxillary premolars on both sides.
* No previous reported or observed dental treatment to the teeth to be extracted.
* No previous reported or observed trauma to the teeth to be extracted.
* No previous reported or observed orthodontic treatment involving the teeth to be extracted.
* Free of any systemic disease affecting the dentition.

Exclusion Criteria:

* Past or present signs or symptoms of periodontal disease.
* Past or present signs or symptoms of bruxism.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Dentin Phosphoprotein levels | 2 months
  Evaluate and compare the possible effect of continuous and intermittent orthodontic forces on root resorption using dentin phosphoprotein levels.

CONTACTS AND LOCATIONS:
Overall Officials: sherifa ghaleb, Principal Investigator — Alexandria University
Locations (2):
- Egypt (2):
  - Faculty of Dentistry,Alexandria University, Alexandria, Please Select A Region, State Or Province.
  - Faculty of Dentistry, Alexandria University, Alexandria

IPD SHARING:
Plan to Share IPD: Yes
Age, Gender
Supporting Information: Study Protocol
Time Frame: 6 months after any publication.
Access Criteria: It will be accessible to all

REFERENCES:
- [Derived] Ghaleb S, Tamish N, ElKenany W, Guindi M. The effect of two different types of forces on possible root resorption in relation to dentin phosphoprotein levels: a single-blind, split-mouth, randomized controlled trial. Prog Orthod. 2021 Dec 20;22(1):44. doi: 10.1186/s40510-021-00388-y. PMID 34927213